CLINICAL TRIAL: NCT05625984
Title: Multi-centre, Open-label, First-in-man Study With Fascigel Used in Adult Patients Suffered From Back Pain
Brief Title: Study With Fascigel
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Contipro Pharma a.s. (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PT-FAS-1_11-21
Record Dates: First submitted 2022-11-15; First posted 2022-11-23 (Actual); Last update posted 2024-02-07 (Actual); Status verified 2024-02

CONDITIONS: Back Pain
MeSH Terms: conditions — Back Pain

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Fascigel injection application (Experimental): Device is administered injected interfascially in the concerned place (low back) in multiple places laterally.
  Interventions: Device: Fascigel

INTERVENTIONS:
Device: Fascigel — The product is a Class III Medical Device. Structure is made by 1% sodium hyaluronate polysaccharide in normal saline solution.

SUMMARY:
The product is a Class III Medical Device. Structure is made by 1% sodium hyaluronate polysaccharide in normal saline solution. The device intended use is to help treat back pain by lubricating fascia.

ELIGIBILITY:
Inclusion Criteria:

* Back pain (VAS above 4 cm)
* Limited range of motion
* Duration of pain for over 3 months
* Patient willing and able to provide the written consent
* Ability to communicate well with the investigator in the local language, and to understand and comply with the requirements of the study

Exclusion Criteria:

* State after back surgery
* BMI > 35
* Age < 18 years
* Pregnant or lactating woman
* Patient in terminal stage of living
* Patient with known hypersensitivity or allergy to any of substances contained in Medical Device
* Patient participating in the intervention clinical study
* Alcohol or drug abuse
* Patient undergoing chronic coagulation therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2022-10-24 (Actual); Primary Completion 2023-11-13 (Actual); Study Completion 2023-11-13 (Actual)

PRIMARY OUTCOMES:
- Pain management | 3 months
  Visual Analogue Scale - 0-100 - higher scores mean a worse outcome

CONTACTS AND LOCATIONS:
Locations (3):
- Czechia (3):
  - Medicinecare s.r.o., Brno
  - FN Královské Vinohrady, Prague
  - FN Motol, Prague